CLINICAL TRIAL: NCT04188171
Title: Sclerotherapy With Polidocanol Foam In The Management Of First, Second And Third-Grade Hemorrhoidal Disease In Patients With Bleeding Disorders: A Prospective Cohort Study
Brief Title: Sclerotherapy With Polidocanol Foam In The Treatment Of Hemorrhoidal Disease In Patients With Bleeding Disorders
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Paulo Sérgio Durão Salgueiro, Principal Investigator, Universidade do Porto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12422301
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Hemorrhoids; Bleeding Disorder
Keywords: Sclerotherapy; Polidocanol foam; Hemorrhoidal disease
MeSH Terms: conditions — Hemorrhoids; Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective study including adult patients, with or without bleeding disorders, with hemorrhoidal disease grades I to III submitted to polidocanol foam sclerotherapy in three health institutions during an inclusion period of 1.5 years. Efficacy and safety outcomes will be compared between two groups of patients: with bleeding disorders (Group A) and without bleeding disorders (Group B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polidocanol foam sclerotherapy (Experimental): During the intervention period the participants are observed at 3-week intervals (maximum of 3 sessions).
  The required number of polidocanol foam sclerotherapy sessions (maximum of 3) is determined by clinical and anoscopic evaluation (if the participant is non-symptomatic and/or there is no significant hemorrhoidal disease on anoscopy, the patient will not be a candidate for additional instrumental therapy moving directly to the follow-up period). After each session all patients were instructed to adopt dietary measures and adequate hydration maintaining therapy with systemic venotropic, topical and laxative if necessary.
  After the intervention period, a one-year follow-up is scheduled with medical appointments performed every 3 months.
  Interventions: Procedure: Polidocanol foam sclerotherapy

INTERVENTIONS:
Procedure: Polidocanol foam sclerotherapy — * Preparation of the foam is done according to the Tessari technique (2 disposable 20ml syringe, a three-way tap, reusable extender adapted to intravenous needle).
  * Sclerosant applied according to the Blanchard technique through a disposable transparent anoscope (patient in knee-chest position).
  * In each session, treatment can be performed on more than one hemorrhoidal cushion. The maximum dose per treatment session is 20ml (mixture of 4ml of polidocanol 3% with 16ml of air).
  * During the intervention period the participants are observed at 3-week intervals. The required number of sessions (maximum of 3) is determined by clinical and anoscopic evaluation.
  * After the intervention period, a one-year follow-up is scheduled with medical appointments performed every 3 months.

SUMMARY:
Treatment of hemorrhoidal disease includes a conservative approach (dietary and behavioral measures, venotropic and topical medication), office-based treatments and surgery. Rubber banding is currently considered the instrumental method of choice in the treatment of hemorrhoidal disease grades I to III (Goligher's classification). However, its use in patients with bleeding disorders is not recommended. Sclerotherapy can be performed in these patients since the hemorrhagic risk is very low. The most commonly used agent for sclerotherapy is liquid polidocanol. Polidocanol foam seems to be more effective than the liquid formulation and is safe in the treatment of hemorrhoidal disease even in patients with coagulation disorders. This study is aimed to evaluate the efficacy and safety of polidocanol foam sclerotherapy in the treatment of hemorrhoidal disease grades I to III in patients with bleeding disorders.

DETAILED DESCRIPTION:
Internal hemorrhoidal disease is classified according to the Goligher classification into grades I, II, III and IV according to its grade of prolapse and reducibility. The treatment of patients should be oriented by the presence of symptoms and the impact on life quality, aspects that are valued on the Sodergren scale.

The hemorrhoidal bleeding, usually mild, may be severe in patients under antithrombotic medications (antiplatelet or anticoagulant) as well as in patients with bleeding disorders non-induced by drugs. With the increase of life expectancy and the high prevalence of atrial fibrillation, the consumption of anticoagulants has also been increasing. Similarly, the use of antiplatelet medication has also increased, especially through its use in the primary and secondary prevention of cardiovascular events. Vitamin K antagonists and antiplatelet drugs are associated with an incidence of digestive bleeding between 1.5% - 4.5% with a short-term mortality of 10-15%. The relation between the use of new oral anticoagulants (NOACs) and digestive bleeding remains a matter of debate, with some studies showing different results when comparing bleeding risk with vitamin K antagonists. Similar to what happen with this subset of patients, those with inherited bleeding disorders are a known subgroup of patients predisposed to hemorrhagic complications. Hemophilia represents the main cause of inherited defects of clotting factors VIII and IX. With the advent of intravenous clotting factors concentrates, the perioperative mortality in this subgroup as decreased in the mid-20th century. However patients with this hematologic disease still have a higher risk of bleeding, delayed wound healing and postoperative infections. To the investigator's knowledge little is known about the prevalence of hemorrhoidal disease in patients with inherited bleeding disorders. Bearing in mind the high rate of surgical complications in these patients, they could represent the ideal candidates for less invasive office-based hemorrhoidal therapy. Instrumental, office-based treatment is reserved for internal hemorrhoidal disease grades I to III. Regardless of the applied technique, the goal is to decrease vascularization, decrease hemorrhoidal volume and increase the fixation of the fibrovascular pedicle to the rectal wall, thus treating the bleeding and hemorrhoidal prolapse. Rubber band ligation is considered the method of choice in the treatment of hemorrhoidal disease. However, its use is associated to bleeding rates after procedure ranging between 3.5 - 50% and late bleeding rates between 13% - 18,3% that may occur until 7-14 days after treatment. The hemorrhagic event is significant in 0.8% of cases and may even prove fatal. For this reason, this technique is contraindicated in patients with bleeding disorders. In patients on antithrombotic medication, discontinuation of this medication is recommended for 7 days before the ligation procedure and 7-10 days after the procedure, which substantially increases the risk of cardioembolic events. In contrast, sclerotherapy is a technique with a low rate of bleeding complications and can be used to treat hemorrhoidal disease grades I to III. After intravascular injection of sclerosing agent above the pectineal line - Blanchard technique - an inflammatory and fibrotic response is obtained that interrupts the blood supply. Although there are multiple sclerosing agents, in Portugal, the most frequently used is liquid polidocanol. As a nonionic detergent its use as a foam (obtained by the technique of Tessari which uses a device that combines two syringes and a three-way tap in which the polidocanol is mixed with air under mechanical force) appears to be associated with greater efficacy even with lower doses of sclerosing agent. Sclerotherapy with liquid polidocanol is effective in the treatment of grade I hemorrhoidal disease with a study demonstrating superiority of foam formulation in this grade of hemorrhoidal disease. A recently published Portuguese study sought to study the efficacy and safety of foamed polidocanol sclerotherapy in patients with grade I to IV hemorrhoidal disease. On the findings, which included 2000 participants, 210 of them on anticoagulant and/or dual antiplatelet therapy, the authors conclude that this instrumental procedure is effective and safe even in patients on antithrombotic therapy. However, no comparison was made between the incidence of complications occurred in this subgroup of patients with the remaining patients without antithrombotic therapy. As far as we know there are no published studies comparing polidocanol foam sclerotherapy to other ablative techniques.

The investigators are conducting a multicentric longitudinal prospective study including adult patients, with or without bleeding disorders, with hemorrhoidal disease grades I to III submitted to polidocanol foam sclerotherapy in three health institutions during an inclusion period of 1.5 years. Efficacy is assessed using Sodergren score of symptoms, bleeding and Goligher grades, and recurrence during follow-up. For the safety evaluation, complications are recorded. Efficacy and safety outcomes will be compared between two groups of patients: with bleeding disorders (Group A) and without bleeding disorders (Group B).

ELIGIBILITY:
Participants will be recruited from August 1st, 2018 until February 1st, 2020.

Inclusion Criteria:

* Adult patients with symptomatic internal hemorrhoidal disease grades I to III submitted to sclerotherapy with polidocanol foam in three Portuguese health institutions (Centro Hospitalar Universitário do Porto, Hospital Senhora da Oliveira - Guimarães and Hospital Prof. Doutor Fernando da Fonseca, EPE - Amadora);
* Hemorrhoidal disease refractory to conservative therapy (dietary modification, intestinal transit modifiers, topical and venotropic drugs) during a period no less than 4 weeks;

Exclusion Criteria:

* Known allergy to polidocanol;
* Liver cirrhosis;
* Pregnant or lactating women;
* Inflammatory bowel disease;
* Other concomitant symptomatic perianal disease;
* History of office-based or surgical treatment of hemorrhoidal disease in the last 6 months;
* Immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness evaluation (therapeutic success) | 3 months
  For efficacy evaluation during the intervention period the outcomes will be compared between groups A and B.
  Therapeutic success is a compound variable of Sodergren symptom score and bleeding grade and is subdivided in:
  * Complete (Sodergren score = 0 and bleeding grade ≤ 1);
  * Partial (Sodergren score> 0 and bleeding grade> 1 but with improvement over initial score); - Therapeutic failure (participants that, after 3 sessions of office-based treatment worsened or maintained the initial Sodergren score and bleeding grade).
Safety evaluationL occurrence of complications | 12 months
  Comparison of the occurrence of complications in both groups A and B.
  Complications are classified as:
  * Mild (e.g. pain/discomfort, minor bleeding, external hemorrhoidal thrombosis not requiring surgical intervention);
  * Moderate (e.g. external hemorrhoidal thrombosis requiring surgical intervention, moderate bleeding not requiring blood transfusion, urgent hemostasis or urgent surgery);
  * Severe (e.g. sepsis, Fournier's gangrene, perineal abscess, bleeding with hemodynamic instability, transfusional need or urgent surgery, sexual impotence in man).

SECONDARY OUTCOMES:
Effectiveness evaluation (Goligher classification) | 3 months
  For efficacy evaluation during the intervention period the outcomes will be compared between groups A and B.
  Variation of Goligher classification before and after the intervention.
Effectiveness evaluation (number of office-based sessions) | 3 months
  Number of office-based therapy sessions and polidocanol foam dose applied during the intervention period (comparing groups A and B).

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Salgueiro, MD, Principal Investigator — Centro Hospitalar Universitário do Porto
Locations (3):
- Portugal (3):
  - Hospital Prof. Doutor Fernando da Fonseca, EPE, Amadora
  - Hospital Senhora da Oliveira, Guimarães
  - Centro Hospitalar Universitário do Porto, Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Halverson A. Hemorrhoids. Clin Colon Rectal Surg. 2007 May;20(2):77-85. doi: 10.1055/s-2007-977485. PMID 20011381
- [Result] Agbo SP. Surgical management of hemorrhoids. J Surg Tech Case Rep. 2011 Jul;3(2):68-75. doi: 10.4103/2006-8808.92797. PMID 22413048
- [Result] Riss S, Weiser FA, Schwameis K, Riss T, Mittlbock M, Steiner G, Stift A. The prevalence of hemorrhoids in adults. Int J Colorectal Dis. 2012 Feb;27(2):215-20. doi: 10.1007/s00384-011-1316-3. Epub 2011 Sep 20. PMID 21932016
- [Result] Everhart JE, Ruhl CE. Burden of digestive diseases in the United States part II: lower gastrointestinal diseases. Gastroenterology. 2009 Mar;136(3):741-54. doi: 10.1053/j.gastro.2009.01.015. Epub 2009 Jan 21. No abstract available. PMID 19166855
- [Result] Johanson JF, Sonnenberg A. The prevalence of hemorrhoids and chronic constipation. An epidemiologic study. Gastroenterology. 1990 Feb;98(2):380-6. doi: 10.1016/0016-5085(90)90828-o. PMID 2295392
- [Result] Qureshi WA. Office management of hemorrhoids. Am J Gastroenterol. 2018 Jun;113(6):795-798. doi: 10.1038/s41395-018-0020-0. No abstract available. PMID 29487411
- [Result] Pucher PH, Qurashi M, Howell AM, Faiz O, Ziprin P, Darzi A, Sodergren MH. Development and validation of a symptom-based severity score for haemorrhoidal disease: the Sodergren score. Colorectal Dis. 2015 Jul;17(7):612-8. doi: 10.1111/codi.12903. PMID 25603811
- [Result] Pengo V, Pegoraro C, Cucchini U, Iliceto S. Worldwide management of oral anticoagulant therapy: the ISAM study. J Thromb Thrombolysis. 2006 Feb;21(1):73-7. doi: 10.1007/s11239-006-5580-y. PMID 16475046
- [Result] Yusuf S, Islam S, Chow CK, Rangarajan S, Dagenais G, Diaz R, Gupta R, Kelishadi R, Iqbal R, Avezum A, Kruger A, Kutty R, Lanas F, Lisheng L, Wei L, Lopez-Jaramillo P, Oguz A, Rahman O, Swidan H, Yusoff K, Zatonski W, Rosengren A, Teo KK; Prospective Urban Rural Epidemiology (PURE) Study Investigators. Use of secondary prevention drugs for cardiovascular disease in the community in high-income, middle-income, and low-income countries (the PURE Study): a prospective epidemiological survey. Lancet. 2011 Oct 1;378(9798):1231-43. doi: 10.1016/S0140-6736(11)61215-4. Epub 2011 Aug 26. PMID 21872920
- [Result] Sorensen R, Hansen ML, Abildstrom SZ, Hvelplund A, Andersson C, Jorgensen C, Madsen JK, Hansen PR, Kober L, Torp-Pedersen C, Gislason GH. Risk of bleeding in patients with acute myocardial infarction treated with different combinations of aspirin, clopidogrel, and vitamin K antagonists in Denmark: a retrospective analysis of nationwide registry data. Lancet. 2009 Dec 12;374(9706):1967-74. doi: 10.1016/S0140-6736(09)61751-7. PMID 20006130
- [Result] Rothberg MB, Celestin C, Fiore LD, Lawler E, Cook JR. Warfarin plus aspirin after myocardial infarction or the acute coronary syndrome: meta-analysis with estimates of risk and benefit. Ann Intern Med. 2005 Aug 16;143(4):241-50. doi: 10.7326/0003-4819-143-4-200508160-00005. PMID 16103468
- [Result] Holster IL, Valkhoff VE, Kuipers EJ, Tjwa ETTL. New oral anticoagulants increase risk for gastrointestinal bleeding: a systematic review and meta-analysis. Gastroenterology. 2013 Jul;145(1):105-112.e15. doi: 10.1053/j.gastro.2013.02.041. Epub 2013 Mar 5. PMID 23470618
- [Result] He Y, Wong IC, Li X, Anand S, Leung WK, Siu CW, Chan EW. The association between non-vitamin K antagonist oral anticoagulants and gastrointestinal bleeding: a meta-analysis of observational studies. Br J Clin Pharmacol. 2016 Jul;82(1):285-300. doi: 10.1111/bcp.12911. Epub 2016 Apr 15. PMID 26889922
- [Result] Pannach S, Goetze J, Marten S, Schreier T, Tittl L, Beyer-Westendorf J. Management and outcome of gastrointestinal bleeding in patients taking oral anticoagulants or antiplatelet drugs. J Gastroenterol. 2017 Dec;52(12):1211-1220. doi: 10.1007/s00535-017-1320-7. Epub 2017 Feb 16. PMID 28210867
- [Result] Craddock CG Jr, Fenninger LD, Simmons B. Hemophilia: Problem of Surgical Intervention for Accompanying Diseases. Review of the Literature and Report of a Case. Ann Surg. 1948 Nov;128(5):888-903. doi: 10.1097/00000658-194811000-00002. No abstract available. PMID 17859247
- [Result] Ingerslev J, Hvid I. Surgery in hemophilia. The general view: patient selection, timing, and preoperative assessment. Semin Hematol. 2006 Jan;43(1 Suppl 1):S23-6. doi: 10.1053/j.seminhematol.2005.11.024. PMID 16427380
- [Result] Cocorullo G, Tutino R, Falco N, Licari L, Orlando G, Fontana T, Raspanti C, Salamone G, Scerrino G, Gallo G, Trompetto M, Gulotta G. The non-surgical management for hemorrhoidal disease. A systematic review. G Chir. 2017 Jan-Feb;38(1):5-14. doi: 10.11138/gchir/2017.38.1.005. PMID 28460197
- [Result] Cataldo P, Ellis CN, Gregorcyk S, Hyman N, Buie WD, Church J, Cohen J, Fleshner P, Kilkenny J 3rd, Ko C, Levien D, Nelson R, Newstead G, Orsay C, Perry WB, Rakinic J, Shellito P, Strong S, Ternent C, Tjandra J, Whiteford M; Standards Practice Task Force, The American Society of Colon and Rectal Surgeons, USA. Practice parameters for the management of hemorrhoids (revised). Dis Colon Rectum. 2005 Feb;48(2):189-94. doi: 10.1007/s10350-004-0921-4. No abstract available. PMID 15711856
- [Result] Davis BR, Lee-Kong SA, Migaly J, Feingold DL, Steele SR. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Management of Hemorrhoids. Dis Colon Rectum. 2018 Mar;61(3):284-292. doi: 10.1097/DCR.0000000000001030. No abstract available. PMID 29420423
- [Result] Albuquerque A. Rubber band ligation of hemorrhoids: A guide for complications. World J Gastrointest Surg. 2016 Sep 27;8(9):614-620. doi: 10.4240/wjgs.v8.i9.614. PMID 27721924
- [Result] Nelson RS, Ewing BM, Ternent C, Shashidharan M, Blatchford GJ, Thorson AG. Risk of late bleeding following hemorrhoidal banding in patients on antithrombotic prophylaxis. Am J Surg. 2008 Dec;196(6):994-9; discussion 999. doi: 10.1016/j.amjsurg.2008.07.036. PMID 19095121
- [Result] Kim M, Song HJ, Kim S, Cho YK, Kim HU, Song BC, Chang WY, Kim SH. Massive life-threatening lower gastrointestinal hemorrhage caused by an internal hemorrhoid in a patient receiving antiplatelet therapy: a case report. Korean J Gastroenterol. 2012 Oct;60(4):253-7. doi: 10.4166/kjg.2012.60.4.253. PMID 23089912
- [Result] Odelowo OO, Mekasha G, Johnson MA. Massive life-threatening lower gastrointestinal hemorrhage following hemorrhoidal rubber band ligation. J Natl Med Assoc. 2002 Dec;94(12):1089-92. PMID 12510709
- [Result] Patel S, Shahzad G, Rizvon K, Subramani K, Viswanathan P, Mustacchia P. Rectal ulcers and massive bleeding after hemorrhoidal band ligation while on aspirin. World J Clin Cases. 2014 Apr 16;2(4):86-9. doi: 10.12998/wjcc.v2.i4.86. PMID 24749117
- [Result] Madoff RD, Fleshman JW; Clinical Practice Committee, American Gastroenterological Association. American Gastroenterological Association technical review on the diagnosis and treatment of hemorrhoids. Gastroenterology. 2004 May;126(5):1463-73. doi: 10.1053/j.gastro.2004.03.008. No abstract available. PMID 15131807
- [Result] Forlini A, Manzelli A, Quaresima S, Forlini M. Long-term result after rubber band ligation for haemorrhoids. Int J Colorectal Dis. 2009 Sep;24(9):1007-10. doi: 10.1007/s00384-009-0698-y. Epub 2009 Apr 23. PMID 19387663
- [Result] Atallah S, Maharaja GK, Martin-Perez B, Burke JP, Albert MR, Larach SW. Transanal hemorrhoidal dearterialization (THD): a safe procedure for the anticoagulated patient? Tech Coloproctol. 2016 Jul;20(7):461-6. doi: 10.1007/s10151-016-1481-z. Epub 2016 May 12. PMID 27170327
- [Result] Sneider EB, Maykel JA. Diagnosis and management of symptomatic hemorrhoids. Surg Clin North Am. 2010 Feb;90(1):17-32, Table of Contents. doi: 10.1016/j.suc.2009.10.005. PMID 20109630
- [Result] Acheson AG, Scholefield JH. Management of haemorrhoids. BMJ. 2008 Feb 16;336(7640):380-3. doi: 10.1136/bmj.39465.674745.80. No abstract available. PMID 18276714
- [Result] ASGE Technology Committee; Siddiqui UD, Barth BA, Banerjee S, Bhat YM, Chauhan SS, Gottlieb KT, Konda V, Maple JT, Murad FM, Pfau P, Pleskow D, Tokar JL, Wang A, Rodriguez SA. Devices for the endoscopic treatment of hemorrhoids. Gastrointest Endosc. 2014 Jan;79(1):8-14. doi: 10.1016/j.gie.2013.07.021. Epub 2013 Nov 14. PMID 24239254
- [Result] Tessari L, Cavezzi A, Frullini A. Preliminary experience with a new sclerosing foam in the treatment of varicose veins. Dermatol Surg. 2001 Jan;27(1):58-60. PMID 11231246
- [Result] Cavezzi A, Tessari L. Foam sclerotherapy techniques: different gases and methods of preparation, catheter versus direct injection. Phlebology. 2009 Dec;24(6):247-51. doi: 10.1258/phleb.2009.009061. PMID 19952380
- [Result] Nastasa V, Samaras K, Ampatzidis Ch, Karapantsios TD, Trelles MA, Moreno-Moraga J, Smarandache A, Pascu ML. Properties of polidocanol foam in view of its use in sclerotherapy. Int J Pharm. 2015 Jan 30;478(2):588-96. doi: 10.1016/j.ijpharm.2014.11.056. Epub 2014 Nov 26. PMID 25433198
- [Result] Yuksel BC, Armagan H, Berkem H, Yildiz Y, Ozel H, Hengirmen S. Conservative management of hemorrhoids: a comparison of venotonic flavonoid micronized purified flavonoid fraction (MPFF) and sclerotherapy. Surg Today. 2008;38(2):123-9. doi: 10.1007/s00595-007-3582-9. Epub 2008 Feb 1. PMID 18239868
- [Result] Moser KH, Mosch C, Walgenbach M, Bussen DG, Kirsch J, Joos AK, Gliem P, Sauerland S. Efficacy and safety of sclerotherapy with polidocanol foam in comparison with fluid sclerosant in the treatment of first-grade haemorrhoidal disease: a randomised, controlled, single-blind, multicentre trial. Int J Colorectal Dis. 2013 Oct;28(10):1439-47. doi: 10.1007/s00384-013-1729-2. Epub 2013 Jun 18. PMID 23775099
- [Result] Fernandes V, Fonseca J. Polidocanol Foam Injected at High Doses with Intravenous Needle: The (Almost) Perfect Treatment of Symptomatic Internal Hemorrhoids. GE Port J Gastroenterol. 2019 May;26(3):169-175. doi: 10.1159/000492202. Epub 2018 Aug 31. PMID 31192285